CLINICAL TRIAL: NCT06545929
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Phase 2 Study to Evaluate Impact of Sunobinop (V117957) on Alcohol Craving in Subjects Diagnosed With Moderate to Severe Alcohol Use Disorder and Seeking Treatment
Brief Title: Study of Sunobinop on Craving in Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imbrium Therapeutics (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUN2003B
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol craving; Moderate to severe alcohol use disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sunobinop (Experimental)
  Interventions: Drug: Sunobinop
- Placebo to match sunobinop (Placebo Comparator)
  Interventions: Drug: Placebo to match sunobinop

INTERVENTIONS:
Drug: Sunobinop — 1 tablet taken orally at bedtime
  Other Names: V117957
  Arms: Sunobinop
Drug: Placebo to match sunobinop — 1 tablet taken orally at bedtime
  Arms: Placebo to match sunobinop

SUMMARY:
The purpose of this study is to evaluate the efficacy of sunobinop compared to placebo on alcohol craving in subjects with moderate to severe alcohol use disorder and these subjects are seeking treatment.

ELIGIBILITY:
Key Inclusion Criteria include:

* Male and female age ≥18 years.
* Diagnosis of moderate or severe alcohol use disorder.
* Currently seeking treatment for alcohol use disorder.
* Has 4 or more heavy drinking days (HDD) in each of the 4 weeks prior to baseline visit.

Key Exclusion Criteria include:

* Subjects that meet current DSM-5 criteria for moderate or severe substance use disorder other than alcohol and nicotine.

Other protocol-specific inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Alcohol Urge Questionnaire (AUQ) | Day 14
  The questionnaire consists of 8 items; each with 7-item scale in which 1= "strongly disagree" and 7 = "strongly agree".

SECONDARY OUTCOMES:
Desire for Alcohol Visual Analog Scale (DFA-VAS) | Day 14
  The scale consists of 1 item with 10-point scale in which 0 = "not at all" and 10 = "extremely high"

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio Clinical Trials, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No